CLINICAL TRIAL: NCT02062775
Title: A Randomized Controlled Study of Self Fixating Mesh Versus Non Fixating Polyester Mesh for Laparoscopic Inguinal Hernia Repair
Brief Title: Comparison of Self-Fixating vs Non-Fixating Hernia Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EH13-356
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-Fixating Hernia Mesh (Active Comparator): Self-fixating polyester mesh will be used for laparoscopic inguinal hernia repair.
  Interventions: Procedure: Use of self-fixating mesh for inguinal hernia repair; Procedure: Absorbable tacks may be used in hernias >2cm
- Non-Fixating Hernia Mesh (Placebo Comparator): Non-fixating polyester mesh will be used for laparoscopic hernia repair.
  Interventions: Procedure: Use of non-fixating mesh for inguinal hernia repair

INTERVENTIONS:
Procedure: Use of self-fixating mesh for inguinal hernia repair — Parietex ProGrip will be used to repair inguinal hernia
  Other Names: Parietex ProGrip
  Arms: Self-Fixating Hernia Mesh
Procedure: Use of non-fixating mesh for inguinal hernia repair — Parietex Anatomic mesh will be used to repair inguinal hernias.
  Other Names: Parietex Anatomic
  Arms: Non-Fixating Hernia Mesh
Procedure: Absorbable tacks may be used in hernias >2cm — Patients randomized to the Parietex ProGrip study group will be further randomized to either receive absorbable tacks or no tacks if the hernia measures >2cm
  Arms: Self-Fixating Hernia Mesh

SUMMARY:
The purpose of this study is to determine if self-fixating polyester mesh will have lower incidence of chronic postoperative pain and recurrence than non-fixating polyester mesh when used for laparoscopic inguinal hernia repair.

DETAILED DESCRIPTION:
This is a randomized, blinded comparison of self-gripping mesh and standard polyester mesh for laparoscopic, primary inguinal hernia repair performed in a Totally ExtraPeritoneal (TEP) fashion.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* ASA Classification I, II, III
* scheduled for elective TEP inguinal hernia repair

Exclusion Criteria:

* ASA Classification IV or greater
* needing emergency surgery
* known history of narcotic dependence
* undergoing bilateral inguinal or combined umbilical hernia repair
* undergoing other procedures during same anesthetic
* undergoing recurrent inguinal hernia repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2013-08; Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Chronic postoperative pain | 1 year

SECONDARY OUTCOMES:
Incidence of hernia recurrence | 1 year

OTHER OUTCOMES:
Post-Op adverse events related to mesh | 1 year
Post-Op quality of life and pain scores | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Linn, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States